CLINICAL TRIAL: NCT05946057
Title: Patient Registry for Individuals With Otoferlin-Associated Hearing Loss
Brief Title: Otoferlin Patient Registry and Natural History Study
Status: Recruiting | Type: Observational
Sponsor: Tobias Moser (Other)
Responsible Party: Sponsor-Investigator, Tobias Moser, Prof., University Medical Center Goettingen
Organization: University Medical Center Goettingen (Other)
Other Study IDs: 17/8/22 v1.1 - 2023-02528
Record Dates: First submitted 2023-06-05; First posted 2023-07-14 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Otoferlin-related Auditory Synaptopathy; Hearing Impairment
Keywords: Otoferlin patient registry; Natural history study
MeSH Terms: conditions — Hearing Loss | interventions — Audiometry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 25 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Otoferlin participant group: Individuals with hearing impairment who have a molecular genetic diagnosis involving otoferlin
  Interventions: Diagnostic Test: Molecular genetic testing and audiometry

INTERVENTIONS:
Diagnostic Test: Molecular genetic testing and audiometry — Genetic testing and audiometry are the interventions of interest

SUMMARY:
This registry is designed to collect comprehensive information about the molecular genetic diagnoses of individuals with otoferlin-associated hearing impairment and clinical information to support a natural history study.

DETAILED DESCRIPTION:
A patient registry, in both German and English languages, has been established for patients with hereditary hearing impairment due to variants in otoferlin (OTOF). The study is conducted in accordance with the current version of the Declaration of Helsinki. The study protocol and database structure have been approved by the Ethics Committee of the University Medical Center Göttingen.

Main objective criterion:

To increase understanding of natural history, types of genetic variants and to facilitate clinical and basic research on otoferlin-associated hearing impairment.

Secondary objective criterion:

To improve knowledge to better characterize individuals with otoferlin-associated hearing impairment in the long term and create prerequisites for improved, patient tailored therapy and care.

ELIGIBILITY:
Inclusion Criteria:

* A molecular genetic diagnosis involving biallelic variants in otoferlin (OTOF) and audiometry

Exclusion Criteria:

* Patients with evidence of non-OTOF molecular genetic diagnoses

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with hearing impairment who have a molecular geneic diagnosis involving otoferlin
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2048-02-21 (Estimated); Study Completion 2048-02-21 (Estimated)

PRIMARY OUTCOMES:
Pure-tone audiometry | 1 year, year 1, according to participant consent
  Audiological characteristics
Speech audiometry | 1 year, year 1, according to participant consent
  Audiological characteristics

SECONDARY OUTCOMES:
Otoacoustic emission thresholds | 1 year, year 1, according to participant consent
  Electrophysiological characteristics
Auditory brainstem response | 1 year, year 1, according to participant consent
  Electrophysiological characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Moser, MD, Study Director — University Medical Center Goettingen; Bernd Wollnik, MD, Principal Investigator — University Medical Center Goettingen; Nicola Strenzke, MD, Principal Investigator — University Medical Center Goettingen; Barbara Vona, PhD, Principal Investigator — University Medical Center Goettingen
Locations (1):
- University Medical Center Goettingen, Goettigen, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No
Pseudonymized data will be published in publications

REFERENCES:
- [Result] Vona B, Wollnik B, Strenzke N, Moser T. Catching up but still miles behind-a patient registry for otoferlin. Exp Mol Med. 2024 Jun;56(6):1472-1473. doi: 10.1038/s12276-024-01247-6. Epub 2024 Jun 3. No abstract available. PMID 38825639
- See also: Registry website in German — http://www.auditory-neuroscience.uni-goettingen.de/otoferlin_registry.html
- See also: Registry website in English — http://www.auditory-neuroscience.uni-goettingen.de/otoferlin_registry_en.html

DOCUMENTS (1):
  • Study Protocol: Study Protocol: Study Information English (2025-05-17): https://cdn.clinicaltrials.gov/large-docs/57/NCT05946057/Prot_002.pdf